CLINICAL TRIAL: NCT06897813
Title: A Phase I Randomised, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of WD-910 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Wenda Pharma Technology LTD. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: WD-910-001
Record Dates: First submitted 2025-03-04; First posted 2025-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WD-910 Take a fixed dose of WD-910 tablets orally (Experimental)
  Interventions: Drug: WD-910 tablet
- WD-910 Tablets Placebo Take a fixed dose of WD-910 tablets Placebo orally (Experimental)
  Interventions: Drug: WD-910 Tablets Placebo

INTERVENTIONS:
Drug: WD-910 tablet — Administered P.O.
  Arms: WD-910 Take a fixed dose of WD-910 tablets orally
Drug: WD-910 Tablets Placebo — Administered P.O.
  Arms: WD-910 Tablets Placebo Take a fixed dose of WD-910 tablets Placebo orally

SUMMARY:
This is a phase I, randomised, double-blind, placebo-controlled, 3-part study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of WD-910 in in Healthy Participants Detailed

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years (inclusive) at the time of informed consent.
* Body mass index (BMI) between 18 to 32 kg/m2 and male participant with body weight of ≥ 50.0 kg, female participant with body weight ≥ 45.0 kg

Exclusion Criteria:

* Any major surgery within 12 weeks prior to Day 1, or any planned surgery during the study.
* Poor pill swallowing ability

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs) | A single-ascending dose (SAD) study ：up to 1week; multiple-ascending dose (MAD) study and food effect (FE) study : up to2weeks
Number of participants with abnormal lab values | SAD ：up to 1week; MAD and FE : up to2weeks
Single Ascending Dose Cohorts : Cmax | From Day1 to Day3
Single Ascending Dose Cohorts : AUC0-∞ | From Day1 to Day3
Single Ascending Dose Cohorts : Tmax | From Day1 to Day3
Single Ascending Dose Cohorts : t½ | From Day1 to Day3
Multiple Ascending Dose Cohorts: Cmax,ss | Day1 , Day10
Multiple Ascending Dose Cohorts: Cmin,ss | Day1 , Day10
Multiple Ascending Dose Cohorts: Cavg,ss | Day1 , Day10
Multiple Ascending Dose Cohorts: Tmax,ss | Day1 , Day10
Multiple Ascending Dose Cohorts: AUC0-τ | Day1 , Day10
Multiple Ascending Dose Cohorts: t½, | Day1 , Day10
Food Effect Cohorts: Cmax | From Day1 to Day4 ， From Day8 to Day11
Food Effect Cohorts: Tmax | From Day1 to Day4 ， From Day8 to Day11
Food Effect Cohorts: AUC0-t | From Day1 to Day4 ， From Day8 to Day11

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided